CLINICAL TRIAL: NCT04156347
Title: A Phase I Study of Sequestered Transscleral, Controlled-Release Topotecan Delivered From an Episcleral Reservoir in Retinoblastoma Eyes
Brief Title: Topotecan Episcleral Plaque for Treatment of Retinoblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targeted Therapy Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3TRB01
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-04

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I Open Label Study (Experimental): Phase I Single Arm
  Interventions: Drug: Episcleral Topotecan

INTERVENTIONS:
Drug: Episcleral Topotecan — Transscleral Topotecan
  Other Names: Episcleral Topotecan, Transscleral Topotecan, Sustained Release Episcleral Topotecan, Chemoplaque

SUMMARY:
This single-arm, non-randomized, dose escalation phase I clinical trial will assess primarily the safety and secondarily the efficacy of episcleral topotecan in patients with active de novo or recurrent intraocular retinoblastoma in at least one eye following completion of first-line therapy.

DETAILED DESCRIPTION:
Retinoblastoma is the most common pediatric malignant intraocular tumor and originates from the retina. Treatment of eyes with advanced intraocular retinoblastoma remains a challenge. The historic standard of care for patients with unilateral disease is enucleation and for those with bilateral disease, a variety of modalities have been tried. These include radiation therapy, systemic chemotherapy, periocular administration of chemotherapy, selective intra-arterial chemotherapy, and intravitreal chemotherapy. Unfortunately, all of these modalities are associated with significant morbidity and investigators are looking for new ways to treat these patients either with novel directed drug delivery methods or with new less toxic agents. This study will evaluate the safety and efficacy of topotecan delivered directly to the eye using a novel sustained-release topotecan episcleral delivery system (also referred to as a Chemoplaque) in patients with active de novo or recurrent intraocular retinoblastoma in at least one eye following completion of first-line therapy. The study intervention involves the insertion and removal of the Chemoplaque, examinations under anaesthesia (EUAs), visits to clinic to monitor for adverse events throughout, and post plaque removal toxicity evaluation. EUAs, clinic visits and laboratory tests are standard of care for retinoblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants must be < 21 years of age.

Diagnosis and Treatment. Participants must have:

Unilateral Group D or earlier-stage intraocular retinoblastoma in which enucleation is a recommended therapy, with no previous local or systemic therapy for retinoblastoma with intraocular calcium in the tumor-containing eye by ophthalmic ultrasound or neuroimaging.

OR Active residual or recurrent intraocular retinoblastoma in at least one eye following completion of first-line therapy (focal therapy for IIRC Group A eyes, or systemic or intra-arterial chemotherapy).

One eye will be the Study Eye. When participants have two eyes with retinoblastoma, the eye with worst disease or best vision potential will be designated the Study Eye. There will only be one eye per child treated in this Phase I study, since treatment of two eyes would double the systemic dose of drug. The Non-study eye will be treated by standard of care, with only focal therapy during the Study Period, if required.

Must have demonstrated intraocular calcium in the tumor-containing eye by ophthalmic ultrasound or by neuroimaging as part of standard retinoblastoma diagnosis.

Study eye must have vision potential, at least light perception vision in the tumor-bearing eye either with pupil response testing or demonstration of avoidance behavior to light presentation in the affected eye, and no clinical features suggestive of high risk of extraocular extension.

Performance Level: Lansky greater than or equal 50 (<16 years of age); Karnofsky performance scale of >50 (>16 years of age).

Organ Function Requirements:

1. Adequate Bone Marrow Function defined as:

   * Peripheral absolute neutrophil count (ANC) greater than or equal 1000/mm3
   * Platelet count greater than or equal 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 Days prior to enrollment)
   * Hemoglobin greater than or equal 8.0 g/dL at baseline (may receive RBC transfusions)
2. Adequate Renal Function defined as:

   * Creatinine clearance or radioisotope GFR greater than or equal 70ml/min/1.73 m2 or
   * A serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female

   1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5
   1. to < 2 years 0.6 0.6
   2. to < 6 years 0.8 0.8

   6 to < 7 years 1 1

   The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.
3. Adequate Liver Function defined as:

   * Bilirubin (sum of conjugated + unconjugated) less than or equal 1.5 x upper limit of normal (ULN) for age.
   * SGPT (ALT) less than or equal 110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
   * Serum albumin greater than or requal 2 g/dL.
4. Pregnancy prevention. Females of reproductive potential must agree to the use of highly effective contraception during study participation and for an additional 40 days after the end of Episcleral Topotecan administration.
5. Informed consent. All participants and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will also be obtained.

Exclusion Criteria

Disease status. Participants known to have any of the following are excluded:

1. tumor involving the optic nerve rim
2. clinical or EUA evidence of extraocular extension
3. evidence of metastatic retinoblastoma
4. existing neuroimaging showing suspicion of, or definitive, optic nerve . invasion, trilateral retinoblastoma or extra-ocular extension.

Allergy. Participants with reported allergy to topotecan, camptothecin or derivatives thereof are excluded.

Concomitant treatment. Participants who have received chemotherapy, other focal retinoblastoma therapy or any other investigational agent within 3 weeks of Episcleral Topotecan placement are not eligible.

Uncontrolled intercurrent illness. Participants with known uncontrolled intercurrent illness that, in the investigator's opinion, would put the participant at undue risk or limit compliance with the study requirements, are not eligible.

Febrile illness. Participants with clinically significant febrile illness (as determined by the investigator) within one week prior to initiation of protocol therapy are excluded.

Pregnancy and lactation. Females of reproductive potential must have a negative serum pregnancy test within 72 hours prior to initiation of protocol therapy. Due to the unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with the study agents, breastfeeding must be discontinued if the mother is treated on study.

Compliance. Any condition of diagnosis that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with the study instruction, might confound the interpretation of the study results, or put the participant at risk.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of Episcleral Topotecan in participants with retinoblastoma-Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D). | 9 Weeks
  To determine the safety and tolerability of Episcleral Topotecan in participants with retinoblastoma.

SECONDARY OUTCOMES:
To determine systemic exposure by measurement of Topotecan in plasma. | 42 Days
  To characterize the systemic exposure of episcleral topotecan by quantifying topotecan concentration in plasma.
To preliminarily define the antitumor activity as determine by assessments of tumor reponse; | 42 Days
  To preliminarily define the antitumor activity as determine by assessment of tumor response.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No